CLINICAL TRIAL: NCT03887390
Title: Implementation of the Depression Medication Choice Decision Aid in a Canadian Context: A Feasibility Trial
Brief Title: Depression Medication Choice Decision Aid
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: First the study failed to recruit the required sample size. Second, we no longer have acess to the clinics, due to the coronavirus outbreak
Sponsor: Laval University (Other)
Collaborators: Réseau-1 Québec (Unknown); CERSSPL (Unknown)
Responsible Party: Principal Investigator, Annie Leblanc, Associate Professor, Laval University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 120560
Record Dates: First submitted 2019-03-12; First posted 2019-03-25 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Depression
Keywords: Depression; Decision Aid; Shared Decision Making; Primary Care; Comparative Effectiveness Research
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: This is a mixed-method feasibility study centered on a pilot clinical trial in family medicine groups in Quebec, Canada, accompanied by a realistic qualitative evaluation of process.
Masking Description: Patients will be randomly assigned to one of two groups (intervention or usual care) using a computer-generated sequence. Due to the nature of the study, patients, health professionals, and members of the research team cannot be masked to the allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Participants in this arm will receive care as usual.
- Depression Medication Choice (Experimental): Participants in this arm will have the Depression Medication Choice decision aid be made available to their clinician to be used during their clinical encounter.
  Interventions: Behavioral: Depression Medication Choice

INTERVENTIONS:
Behavioral: Depression Medication Choice — The Depression Medication Choice tool is a series of cards emphasizing issues that are important for the patient and the health care professional when choosing antidepressants: weight change, sexual issues, sleep, cost, side effects, and stopping approach. The Depression Medication Choice tool uses clear language and is designed to improve the understanding of patients regarding the different attributes of antidepressants, and for use during clinical encounters.
  Arms: Depression Medication Choice

SUMMARY:
The quality of care for patients facing depression, one of the most prevalent chronic diseases, needs improvement. Despite its high incidence, depression remains sub-optimally managed, particularly in primary care, where most patients suffering from depression receive care. Successfully treated depressive patients can potentially improve their burden of disease and significantly improve their quality of life, but not without the best treatment adapted to their contexts, preferences, and expectations. Clinical research provides essential knowledge for the delivery of quality care which is unfortunately seldom applied in daily practice.

One of the preferred methods for overcoming this lack of quality of care is shared decision making: a collaborative process between a clinician and patient that relies on the consideration of scientific evidence, in addition to the values and preferences of the patient. The use of decision aids supports this process by presenting scientific information in an accessible manner while focusing on patient-centered discussion. We developed and rigorously evaluated, in the United States, a decision aid regarding pharmaceutical treatment options for depression, Depression Medication Choice, to be used by health professionals and patients during clinical encounters. The integration and impact of Depression Medication Choice, in primary care practices in a Canadian context is unknown.

The specific objectives of this study are threefold: (i) Evaluate the potential impact of the use of Depression Medication Choice by health professionals and patients during clinical encounters on measures of the quality of the decisional process and on health issues important to the patient and health professional; (ii) Document the processes and optimal measures to take to successfully realize projects on a larger scale; and (iii) Evaluate the feasibility of performing patient-centered studies in a realistic context, minimally disturbing to the study environment, in the primary care context in Quebec, Canada.

Once completed, the estimated potential impact of this decision aid and shared decision making in primary care in a Canadian context will have been measured, progressing toward high-quality patient-centered care. Moreover, it will be possible to optimally perform future studies in realistic contexts while minimizing the burden on the clinics, their health professionals, and their patients.

ELIGIBILITY:
Inclusion Criteria:

* Already have or receive a depression diagnosis (according to the treating clinician)
* Speak English of French
* Have no major obstacles providing clear written consent
* Discuss the possibility of taking antidepressants during the clinical encounter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-07-22 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
Changes in decisional conflict assessed by the Decisional Conflict Scale (DCS) | Immediately following each participant's first clinical encounter and every subsequent scheduled visit for the approximate 6-month study intervention duration
  Participants and clinicians will complete a Decisional Conflict Scale so that their level of decisional conflict may be measured. This measure, validated in French, comprises 16-items grouped into factors impacting the feeling of comfort toward making the decision. Scores range from 0 (no decisional conflict) to 100 (extremely high decisional conflict). A participant version as well as a clinician version of the DCS will be used.

SECONDARY OUTCOMES:
Participant engagement assessed by the Observing Patient Involvement in Decision Making instrument (OPTION) and video recordings | At each participant's scheduled clinical encounter, for up to 6 months post-recruitment
  The level to which the clinicians engage the participants in decision making will be evaluated via the 12-item OPTION scale, an observational measurement scored 0 to 100 percent. Independent reviewers will assess the level of engagement using video recordings of the clinical encounters.
Changes in severity of symptoms assessed by the Patient Health Questionnaire (PHQ-9) | Immediately prior to each participant's first clinical encounter and every subsequent scheduled visit for the approximate 6-month study intervention duration
  Participants will complete the PHQ-9, a severity of depression measurement using a 4-point Likert-type scale. Scores range between 0 and 27 and correspond to depression severity. Depression severity may be: none-minimal (0 to 4), mild (5 to 9), moderate (10-14), moderately severe (15-19), or severe (20-27).
Decision making preference assessed by questionnaire | Immediately prior to each participant's first clinical encounter
  Participants will be asked to answer a single question with a 5-point Likert-type scale to rate their decision making preferences. Lower values indicate participants' preference for making decisions themselves while higher values indicate a preference for their doctor to make the decision for them. An intermediate value indicates participants' preference for shared decision making.
Global quality of life assessed by questionnaire | Immediately prior to the first clinical encounter
  Participants will be asked to answer a single question with a 10-point Likert-type scale to rate their quality of life. The question is scored from 1 (very bad) to 10 (very good).
Changes in medication adherence assessed by participants' pharmacy records | Following the approximate 6-month study intervention completion
  The following data will be extracted for the duration of trial participation: new prescriptions filled and the associated renewal dates as well as the types of medication (depression-related).
Fidelity to the intervention delivery | The entire duration of the discussion between the clinician and participant regarding depression medication during each scheduled visit for the approximate 6-month study intervention duration
  Independent reviewers will evaluate the fidelity with which the Depression Medication Choice tool is used during the clinical encounters via video observation. The control of fidelity list is specific to the Depression Medication Choice tool. This will also allow us to validate the contamination level of the clinicians who will navigate between both groups.
Changes in knowledge assessed by questionnaire | Immediately following each participant's clinical encounter and every subsequent visit for the approximate 6-month study intervention duration
  Participants will be asked to complete a questionnaire assessing their knowledge of the illness (depression) and the advantages and disadvantages of 15 pharmacological treatments. Participants may choose to answer true, false, or unsure. Correct answeres are are given a score of 1 and incorrect answers (or if a participant answered "unsure") is given a score of 0. A mean knowledge score is calculated from the totaled items for comparison.
Changes in satisfaction and acceptability by questionnaire | Immediately following the first clinical encounter and every subsequent visit for the approximate 6-month study intervention duration
  Participants and clinicians will be asked to rate their level of satisfaction and acceptability of the decision aid by completing a 5-question questionnaire. The 7-point Likert-type scale is scored from 5 to 35 with higher values corresponding to higher levels of satisfaction and acceptability.

CONTACTS AND LOCATIONS:
Overall Officials: Annie LeBlanc, PhD, Principal Investigator — Laval University
Locations (1):
- Groupe de médecine de famille universitaire Maizerets, Québec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] LeBlanc A, Herrin J, Williams MD, Inselman JW, Branda ME, Shah ND, Heim EM, Dick SR, Linzer M, Boehm DH, Dall-Winther KM, Matthews MR, Yost KJ, Shepel KK, Montori VM. Shared Decision Making for Antidepressants in Primary Care: A Cluster Randomized Trial. JAMA Intern Med. 2015 Nov;175(11):1761-70. doi: 10.1001/jamainternmed.2015.5214. PMID 26414670